CLINICAL TRIAL: NCT06326294
Title: A Randomized Clinical Trial to Assess the Effectiveness of Thermal Ablation Versus Loop Electrosurgical Excision Procedure for Cervical Cancer Risk Reduction in Women Living With Human Immunodeficiency Virus in Mozambique
Brief Title: Assessment of the Effectiveness of TA Versus LEEP for Cervical Cancer Risk Reduction in WLHIV in Mozambique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Saúde, Mozambique (Other Government)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 727/CNBS/23
Record Dates: First submitted 2024-02-27; First posted 2024-03-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections; HPV Infection; CIN 2/3
MeSH Terms: conditions — HIV Infections; Papillomavirus Infections | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Intervention Model Description: To compare TA, an ablative cervical treatment modality, and LEEP, an excisional cervical treatment modality, in screen-positive WLWH patients, for eradication of hrHPV and effectiveness of treating biopsy-confirmed CIN 2/3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thermo ablation treatment (Other): Participants allocated in this group will be treated with thermo ablation. Before TA, perform biopsies of any acetowhite lesions by colposcopy and/or positive by AVE and an endocervical curettage (ECC); In women who do not have any lesions noted by colposcopy or AVE, one random cervical biopsy at the squamocolumnar junction and an endocervical curettage (ECC) will be obtained.
  TA is performed during the same exam (immediately following biopsies/ECC)TA will be done according to the manufacturer's instructions and specifications.
  Interventions: Device: Thermal ablation
- LEEP treatment (Other): Participants allocated in this group will be treated with LEEP. LEEP will be done according to standard procedure. No biopsies are taken, only LEEP is performed, unless clinically indicated.
  Interventions: Procedure: LOOP ELECTROSURGICAL EXCISION PROCEDURE

INTERVENTIONS:
Device: Thermal ablation — Thermal ablative uses heat (100°C to 120°C) to cause localized tissue damage at the cervical transformation zone and destroy the abnormal epithelium.
  Other Names: TA
  Arms: Thermo ablation treatment
Procedure: LOOP ELECTROSURGICAL EXCISION PROCEDURE — Cervical tissue excision
  Other Names: LEEP
  Arms: LEEP treatment

SUMMARY:
Given that WLWH are more likely to develop persistent HPV infection and CC, effective screening and the management and treatment of pre-cancerous cervical abnormalities is critical to decrease the global burden of cervical cancer. The vast majority of WLWH live in SSA, where resources are more constrained. Therefore, simple, affordable, and effective tools are needed for the prevention of cervical cancer in SSA. In this setting, the best method for treatment of screen-positive WLWH has not been determined. The proposed study will compare the effectiveness of TA vs. LEEP, for treating precursor lesions (CIN 2/3) and HPV infection in WLWH, identify the determinants of treatment failure, and develop a strategy to predict patients in whom treatment is likely to fail so that alternative treatments can be provided. Moreover, local evidence of the optimal method of treatments is necessary to inform health policy and promote adherence.

DETAILED DESCRIPTION:
A. General purpose:

The goal of this study is to compare TA, an ablative cervical treatment modality, and LEEP, an excisional cervical treatment modality, in screen-positive WLWH patients, for eradication of hrHPV and effectiveness of treating biopsy-confirmed CIN 2/3.

B. Specific purposes

Primary Objectives:

1. Compare the effectiveness of treating biopsy-confirmed CIN 2/3 by TA versus LEEP
2. Compare the effectiveness of treating hrHPV infection by TA versus LEEP
3. Assess pain and side effects/adverse events due to TA versus LEEP

Secondary Objectives:

1. Identify the determinants of treatment failures
2. Develop a deep learning-based automated visual evaluation tool that predicts treatment failure

ELIGIBILITY:
Inclusion Criteria:

* ages 25-49 years;
* confirmed HIV infection;
* physically and mentally willing and able to participate in the study, and provide informed consent.

Exclusion Criteria:

* currently pregnant or <6 weeks post-partum;
* had a hysterectomy and no longer have a cervix;
* a history of cervical cancer or treatment for cervical abnormalities; and
* any medical, psychiatric, or other condition that would interfere with protocol adherence, assessment of safety, and/or ability/competence to provide informed consent.

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4844 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of treatment success rates for biopsy-confirmed CIN 2/3: Thermoablation (TA) vs. Loop Electrosurgical Excision Procedure (LEEP) | 12 months
  The treatment success rate (12-month efficacy) of LEEP (pL) and that of ablation (pA) for participants with ablation-eligible CIN 2/3 will be measured by assessing the proportion of patients in each treatment group whose lesions completely regress or are successfully treated without recurrence over a defined follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Edna Viegas, MD, PhD, Principal Investigator — Instituto Nacional de Saúde, Mozambique
Locations (1):
- INSMozambique, Maputo, Mozambique

REFERENCES:
- [Derived] Fallah PN, Salcedo MP, Nhacule E, Utui Y, Massinga MM, Osman NB, Tivir GG, Carrilho C, Monteiro E, Rangeiro R, Neves A, Changule D, Mariano A, Machaze A, Castiano CE, Baker E, Jeronimo J, Chiao EY, Munsell MF, Varon ML, Milan J, Thomas JP, Richards-Kortum R, Lorenzoni C, Omar Viegas EN, Castle PE, Schmeler KM. A randomized clinical trial to assess the effectiveness of thermal ablation versus loop electrosurgical excision procedure for cervical cancer risk reduction in women living with HIV in Mozambique. Int J Gynecol Cancer. 2026 Jan;36(1):101905. doi: 10.1016/j.ijgc.2025.101905. Epub 2025 Apr 26. PMID 40399211